CLINICAL TRIAL: NCT04884971
Title: Microbiota Transplant Therapy for Pulmonary Arterial Hypertension: Early Safety and Feasibility Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-2021-29604
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Microbiota Treatment Arm (Experimental): Participants will receive the encapsulated microbiota intervention daily for seven days and will be subsequently monitored for six months.
  Interventions: Drug: Intestinal microbiota transplant (IMT)

INTERVENTIONS:
Drug: Intestinal microbiota transplant (IMT) — Two size 00 capsules from a single lot will be taken daily. Approximately 2.0 x 10^11 bacteria from a healthy donor are contained in each capsule.

SUMMARY:
This pilot clinical trial will evaluate the initial safety and feasibility of intestinal microbiota transplantation (IMT) in patients with pulmonary arterial hypertension (PAH). This trial will inform development of future trials in treatment of PAH. Active drug in capsule form composed of freeze-dried, encapsulated intestinal microbiota from healthy donors will be administered to patients with PAH. This study will also allow for limited evaluation of pharmacokinetics in terms of donor microbiota engraftment and pharmacodynamics in terms of potential mechanisms. It will also allow for limited evaluation of cardiac endurance and function prior to and after IMT.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a chronic disease characterized by pulmonary vascular remodeling of precapillary pulmonary arteries resulting in obstruction, increased pulmonary vascular resistance, right-sided cardiac failure, and ultimately death. Although pharmacologic therapies have been developed, these modestly improve cardiac function and primarily act to improve symptoms and quality of life; therefore, PAH remains a very lethal disease. Perivascular lung inflammation drives these vascular changes in PAH. This inflammatory profile could be driven by an imbalance of pro- and anti-inflammatory intestinal microbial metabolites, cytokines, other mediators, and/or direct effects of circulating bacteria all stemming from dysbiosis, gut-barrier dysfunction, and possibly, decreased hepatic filtration. Because PAH is characterized by a microbiome distinct from healthy controls, the investigators hypothesize that intestinal microbiota transplant (IMT) will help to reduce severity of PAH and improve quality of life, and that the healthy microbiome may exert these effects by decreasing inflammation. In this pilot clinical trial, the investigators aim to test the safety and feasibility of IMT from healthy donors into patients with PAH. Additionally, in the exploratory objectives, the investigators will obtain limited data to study pharmacokinetics of IMT, including engraftment and stability of donor intestinal microbiota, and pharmacodynamics to include circulating microbial products and markers of inflammation. Proposed circulating markers that may be assessed include interleukin-6, C-reactive protein, soluble CD14, lipopolysaccharide (LPS), phenylacetylglutamine, trimethylamine N-oxide, intestinal fatty acid binding protein, zonulin, claudin, short-chain fatty acids (SCFAs), tumor necrosis factor-α, interleukin-1β, and transforming growth factor-β.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulmonary arterial hypertension (PAH)
* On stable treatment for PAH for one month prior to enrollment
* Able to swallow capsultes
* Able to provide blood sample and fecal sample

Exclusion Criteria:

* Dysphagia to pills
* Clinically active inflammatory bowel disease
* Pregnancy or breastfeeding
* Life expectancy of <6 months
* Presence of ileostomy or colostomy
* Taking immunosuppressants (calcineurin inhibitors, prednisone greater than or equal to 20mg/day, methotrexate, azathioprine, immunosuppressive biologics, JAK inhibitors)
* Neurotropenia (an absolute neurotrophil count < 0.5 x 10^9 cells/L)
* History of solid organ or bone marrow transplant
* Anticipated recurrent antibiotic use (participants with frequent urinary tract infections or sinusitis)
* History of severe anaphylactic food allergy
* History of celiac disease
* History of receiving cancer chemotherapy, immunotherapy, or radiation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of Serious Adverse Events | 6 months
  In order to assess the safety of the trial, the frequency of adverse events will be reported. Outcome will be reported as the mean number of serious adverse events per participant.
Proportion of IMT Compliance | 6 months
  In order to assess the feasibility of the trial, the proportion of subjects taking 100% of the intestinal microbiota transplantation (IMT) doses per protocol will be reported. Outcome is reported as the percent of participants who consume 100% of IMT doses.

CONTACTS AND LOCATIONS:
Overall Officials: Thenappan Thenappan, MD, Principal Investigator — University of Minnesota Division of Cardiology; Kurt Prins, MD, PhD, Principal Investigator — University of Minnesota Division of Cardiology; Edward Weir, MD, Principal Investigator — University of Minnesota Division of Cardiology; Alexander Khoruts, MD, Principal Investigator — University of Minnesota Division of Gastroenterology
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moutsoglou D, Blake M, Belhasan DC, Peichel G, Vang BM, Weir EK, Lopez S, Prins KW, Kabage AJ, Prisco SZ, Kremer BP, Khoruts A, Thenappan T. Microbiota Transplant Therapy Is Safe and Feasible in Pulmonary Arterial Hypertension. JACC Basic Transl Sci. 2025 Sep;10(9):101347. doi: 10.1016/j.jacbts.2025.101347. Epub 2025 Aug 12. PMID 40803054